CLINICAL TRIAL: NCT04463966
Title: Tranexamic Acid for the Prevention of Postpartum Haemorrhage
Brief Title: Prevention of Postpartum Haemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Dr. Abou Bakr Mohamed El Nashaar, professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Tranexamic
Record Dates: First submitted 2020-04-30; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Post Partum Hemorrhage
Keywords: tranexamic acid; postpartum hemorrhage; cesarean section
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Active Comparator): Tranexamic acid 1 gm (100 mg/ml) slowly intravenous infusion during delivery ( administered over 10 minutes at 1 ml/minute) .
  Interventions: Drug: Tranexamic acid injection
- Control (No Intervention): control group will not be given tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid injection — 1 gm (100 mg/ml) slowly intravenous infusion during delivery ( administered over 10 minutes at 1 ml/minute) .
  Other Names: Kapron, 500 mg/5ml
  Arms: Study

SUMMARY:
Use of Tranexamic Acid for prevention of Postpartum hemorrhage in high risk patients: Randomized Control Trial

DETAILED DESCRIPTION:
This study aims to assess the efficacy of administration of Tranexamic Acid in preventing Postpartum haemorrhage & reducing intraoperative and postoperative blood loss in high risk women for Postpartum Hemorrhage undergoing caesarean section. Studying its benefit to transfusion-sparing and hysterectomy-sparing. & reduction of hemorrhage-related mortality when Postpartum hemorrhage is expected.

ELIGIBILITY:
Inclusion Criteria:

* Women at high risk for postpartum hemorrhage after cesarean section

Exclusion Criteria:

* women who are not at high risk for postpartum hemorrhage , or attending for normal vaginal delivery.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
blood loss | immediately after deliver
  Estimation of blood loss

SECONDARY OUTCOMES:
blood pressure | immediately after delivery
  blood pressure
pulse | immediately after delivery
  pulse
temperature | immeditely after delivery
  temperature

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa Ezzat, Principal Investigator — Police Hospital
Locations (1):
- Police Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided